CLINICAL TRIAL: NCT00586794
Title: Therapy of Pulmonary Arterial Hypertension (PAH) - Treatment With Sildenafil in Eisenmenger Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Dr. Siegrun Mebus, DHZB,German Heart Institute Munich, Competence Network for Congenital Heart Defects,
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MP 3.1 Sildenafil
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2010-10

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Hypertension; Eisenmenger
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension; Eisenmenger Complex | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Sildenafil
- B (Placebo Comparator): from the 26th weeks on open-label, all patients were treated with Sildenafil
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — 3x per day 20 mg TID
  Other Names: Revatio®
  Arms: A
Drug: Placebo — 3x per day, 20 mg TID
  Arms: B

SUMMARY:
Eisenmenger's syndrome presents as a severe clinical picture of polymorbidity that constitutes a great burden at the individual as well as the familial and social level. The combination of critically increased pulmonary vascular resistance, progressive pressure load of the right ventricle and disturbance of pulmonary gas exchange result in long-term polymorbidity. The objective of this study is to provide evidence of improvement of patients exercise tolerance as well as general conditions by treatment with oral sildenafil as a specific pulmonary vasodilator.

DETAILED DESCRIPTION:
Eisenmenger's syndrome presents as a severe clinical picture of polymorbidity that constitutes a great burden at the individual as well as the familial and social level. The combination of critically increased pulmonary vascular resistance, progressive pressure load of the right ventricle and disturbance of pulmonary gas exchange result in long-term polymorbidity. While the patient's ability to care for him-/ herself gets lost over time, the financial burden due to the need for medical consultations and hospital stays increases. This is distressing to both the patient and the family. Usually, death results from cardiac decompensation in the presence of gradually increasing pulmonary vascular resistance and hypoxic lesion of organs including the myocardium (Hopkins, AJC 2002).

With a better understanding of the pathophysiology underlying pulmonary hypertension, novel therapeutic approaches have been developed during the past few years. These include a) inhibition of the NO-cGMP-degrading type 5 phosphodiesterase (PDE-5) and b) antagonising the endothelin system (Krum, Curr Opin Investig Drugs 2003). The goal is a dilatation of the abnormally constricted pulmonary arterial vessels by relaxation of the vascular smooth muscle cells with a reversal of pulmonary vascular remodelling (Ghofrani, Pneumologie 2002).

Specific drugs affecting pulmonary vascular resistance have been studied. Intravenous prostacyclin has major disadvantages: high cost, tachyphylaxis, risk of infection and rebound hypertension upon discontinuation. Inhalative pulmonary vasodilators, in particular iloprost, may be effective in primary pulmonary hypertension (Olschewski, Ann Int Med 1996; Hoeper, Pneumologie 2001), but administration is time-consuming, and due to its mode of application its effects are intermittent, lasting only about 75 minutes (Hoeper, JACC 2000). Considering this, oral treatments appear preferable, because of easy administration and, hence, better patient compliance.

Sildenafil (Revatio®) an inhibitor of the phosphodiesterase 5 (PDE-5) was used in many individual cases (Abrams, Schulze-Neick et al, Heart 2000), some acute studies and two long-term studies in humans to reduce the pulmonary vessel resistance. Significant effects on reduction of the pulmonary vessel resistance were demonstrated for the combination with an inhalational prostanoid (Ghofrani et al, Ann Int Med 2002).Good long-term tolerability and effectiveness over a period of two year were demonstrated by this working group.

The objective of this study is to provide evidence of improvement of patients exercise tolerance as well as general conditions by treatment with oral sildenafil as a specific pulmonary vasodilator. The data obtained are supposed to contribute to the development of guidelines for the treatment of Pulmonary Arterial Hypertension (PAH)caused by congenital heart defects.

The hypotheses are:

1. Sildenafil heales specific pulmonary vascular damage, which occurs by hypercirculation as quick-acting inhibiting vasoconstriction.
2. Through this there will be a reduction of pulmonary vessel resistance and a normalization of pulmonary reagibility in patients with Eisenmenger syndrome.
3. Pulmonary blood circulation and so systemic arterial oxygen delivery will increase.
4. The patient benefits from this by improving his exercise tolerance as well as general and clinical condition.

These hypotheses will be tested by comparing findings of the following examinations before, during and after the 52 or 78-week treatment with sildenafil: clinical examination, Electrocardiogram (ECG), echocardiography, ergospirometry, Magnetic Resonance Imaging (MRI), cardiac catheterization with pulmonary artery manometry, and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

Non-specific:

1. Written informed consent obtained.
2. No participation in another AMG driven study attendancing this treatment protocol

Specific:

1. Age at least 14 years
2. Presence of cyanosis with < 93 % arterial oxygen saturation (measured by transcutaneous pulse oximetry)
3. Clinical indication for the invasive diagnostic procedures planned for the study is given; this is evaluated on the basis of observation before, during and after medicinal therapy)
4. Presence of PAH as diagnosed by invasive methods with Rp:Rs > 0.5 measured at rest, before testing of pulmonary vasodilatory reserve
5. One of the following diagnoses:

   1. non-corrected large congenital shunting defect at atrial, ventricular or arterial level:

      * PAPVD
      * ASD
      * SVD
      * VSD
      * AVSD
      * TAC
      * APW
      * PDA
      * combinations thereof.
   2. Surgically corrected shunting defect (diagnoses as above) with significant residual defect
   3. Other diagnoses with univentricular physiology/ hemodynamics.

Exclusion Criteria:

Non-specific:

1. pregnancy or lactation
2. women of child-bearing age who are sexually active without practising highly effective methods of contraception
3. any diseases or impairment that, in the opinion of the investigator exclude a subject from participation
4. substance abuse (alcohol, medicines, drugs)
5. other medical, psychological or social circumstances that would adversely affect a patient's ability to participate reliably in the study or increase the risk to themselves or others if they participated
6. insufficient compliance
7. missing willingness to storaging and transferring pseudonymous disease data within this study.
8. subjects who are not able to perform Cardio-Pulmonary Exercise Testing (CPX).

Specific:

1. pulmonary hypertension secondary to any etiology other than those specified in the inclusion criteria
2. subjects with known intolerance of NO and iloprost or their constituents
3. acute decompensated heart failure within the 7 days before the invasive diagnostic procedure
4. clinically significant haemoptysis within the last 6 months
5. hemodynamic instability which would represent an unjustifiable risk during testing of pulmonary arterial vasoreagibility
6. arterial hypotension (as defined by age-specific values)
7. anemia (Hb < 10 g/dl)
8. decompensated symptomatic policythemia; (details: 4.2.2. exclusion criteria)
9. thrombocytopenia (< 50.000/µl)
10. secondary impairment of organic function:

    * impairment of renal function (GFR < 30 ml/min/1,73 m2 BSA)
    * impairment of hepatic function (ALT and/or AST > 3 x ULN and bilirubin ≥ 2 mg/dl)
11. other sources of pulmonary blood flow which prohibit measurement of the blood flow into the lungs and therefore of the pulmonary vascular resistance:

    * Glenn
    * BT shunt
    * significant number of MAPCAs; (details: 4.2.2. exclusion criteria)
12. Obstruction of pulmonary blood outflow:

    * obstruction of pulmonary venous return
    * mitral valve dysfunction
13. Left heart diseases:

    * aortic or mitral valve disease (more severe than "mild")
    * restrictive or congestive cardiomyopathy
    * PCWP/LVEDP > 15 mmHg
    * symptomatic coronary artery disease
14. Significant valvular diseases other than tricuspid or pulmonary regurgitation (these are not exclusion criteria; details: 4.2.2. exclusion criteria).
15. Pericardial constriction
16. History of stroke, myocardial infarction or life-threatening arrhythmia within the 6 months before screening
17. Bronchopulmonary dysplasia (BPD) and other chronic lung diseases
18. History of significant pulmonary embolism
19. Other relevant diseases (e.g. HIV, diabetes mellitus requiring medical treatment)
20. Subjects with trisomy 21 (reproducibility of 6-MWT and CPX doubtful; communication as to side effects and subjective quality of life doubtful)
21. all contraindications against the study medication (see also "4.2.3 concomitant medication")

    * hypersensitivity against the active ingredients as well as supplementaries
    * patients who lost vision on one eye due to a non arteriitic anterior ischaemic neuropathy of the opticus (NAION).

Prohibited concomitant medication:

Any medication listed below which has not been discontinued at least 30 days prior to screening. Specific pulmonary vasodilators during cardiac catheterization are allowed.

1. Unspecified concomitant medication
2. Other significant medication (a.o. chronic intake of systemic immunosuppression as e.g. systemic glucocorticoids, cytostatic drugs, ciclosporin)
3. Instable medication (details: 4.2.5 prohibited concomitant medication):

   * begin of a new medication regimen within the last 30 days before screening
   * change in the dosage of existing medication within the last 7 days before cardiac catheterization
4. Existing anti-pulmonary hypertensive medication (in any form) with:

   * PDE-5 antagonists (e.g. sildenafil)
   * prostanoids (e.g. iloprost, prostacyclin, beraprost) In case the patient is stable and on Bosentan therapy at least for 6 months. Bosentan (Tracleer®) is unprohibited as concomitant medication.
5. Other medication with vascular action:

   * alpha blockers
   * L-arginin (acts through NO axis)
   * ritonavir, nicorandil (act through K+ channels)
6. Medication that is not compatible with sildenafil or interferes with the metabolism:

   * cytochrome P450-CYP2C9 and CYP3A4 inhibitors (e.g. erythromycin/ketoconazole/itraconazole/protease inhibitors)
   * any existing medication that, in the opinion of the investigator, may interfere with sildenafil treatment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
To determine the distance of walking, which is performed during a 6- min walking test; oxygen saturation and relation of resistance Rp : Rs during the examination with "Herzkatheter", described as the difference between visit 1 (baseline) and visit 4 | visit 1 and visit 4 (after 26 weeks)

SECONDARY OUTCOMES:
To provide normalization of pulmonary vascular function (reagibility and vasoactive mediators) in dependence on duration of the therapy | 78 weeks
Parameters of MRI and Echo-diagnostic | 78 weeks
Quality of life (SF-36) | 78 weeks
Safety and tolerance of the treatment | 78 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Siegrun Mebus, MD, Principal Investigator — German Heart Institute Munich, Competence Network for Congenital Heart Defects; Ingram Schulze-Neick, MD, Study Chair — Great Ormond Street Hospital for Sick Children,London
Locations (20):
- Germany (20):
  - Universitätsklinikum Freiburg, Klinik III Päd. Kardiologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum der Universität Heidelberg, Pädiatrische Kardiologie, Heidelberg, Baden-Wurttemberg
  - Medizinische Klinik und Poliklinik, Abteilung Innere Medizin III, Heidelberg, Baden-Wurttemberg
  - Klinikum Stuttgart, Olgahospital, Klinik für Kinderheilkunde und Jugendmedizin, Pädiatrie 3, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Klinik für Kinderheilkunde und Jugendmedizin, Tübingen, Baden-Wurttemberg
  - Deutsches Herzzentrum München, Munich, Bavaria
  - Ludwig-Maximilian-Universität München, Klinikum Großhadern, Abt. Kinderkardiologie und Intensivmedizin, München-Großhadern, Bavaria
  - Universitätsklinikum Giessen and Marburg, Zentrum für Kinderheilkunde und Jugendmedizin, Giessen, Hesse
  - Medizinische Hochschule Hannover, Abt. für Kardiologie und Angiologie, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Klinik für Kinderheilkunde, Pädiatrische Kardiologie und Pädiatrische Intensivmedizin, Hanover, Lower Saxony
  - Elisabeth Kinderkrankenhaus, Zentrum für Kinder- und Jugendmedizin, Oldenburg, Lower Saxony
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Evangelisches und Johanniter Klinikum Niederrhein gGmbH, Herzzentrum Duisburg, Duisburg, North Rhine-Westphalia
  - Universitätsklinikum Münster, EMAH-Zentrum, Münster, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - Universitätsklinikum der Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Charite, Campus Virchow-Klinikum, Otto-Heubner-Centrum für Kinder- und Jugendmedizin, Berlin, State of Berlin
  - Deutsches Herzzentrum Berlin, Abt. angeborener Herzfehler/Kinderkardiologie, Berlin
  - Universitätsklinikum Erlangen, Kinderkardiologische Abteilung, Kinder- und Jugendklinik, Erlangen

REFERENCES:
- See also: (Competence Network for Congenital Heart Defects) — http://www.kompetenznetz-ahf.de